CLINICAL TRIAL: NCT07350915
Title: Randomized Study of Healthy Lifestyle Promotion Using an App Versus Health Education in Sedentary Individuals or Participants in Walking Groups Aged 60 to 80
Brief Title: ActivE³ - Everyone, Everywhere, Everyday WP 2 - Personalized Data-driven Coaching Platform for Stimulating and Promoting Active Lifestyle and Health Risk Prevention
Acronym: Active3-WP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Giuseppe Andreoni, Full Professor, Politecnico di Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Active3-WP2
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): DTx adopters.
  Interventions: Device: Digital Therapeutics
- Control Group (No Intervention): Administered with only standard educational program

INTERVENTIONS:
Device: Digital Therapeutics — coaching App for the promotion of physical activity and balanced nutrition based on Mediterranean diet scheme as a prevention tool for healthy ageing in the 60-80 age group.
  Arms: Intervention Group

SUMMARY:
The objective of WP2 of the Active3 project is to develop a digital solution for promoting and monitoring physical activity in social settings (real or virtual) that implements a Preventive Medicine approach to healthy aging.

Specifically, the objective of the action related to Word Package 2 is to develop a personalized, data-driven coaching platform co-designed with local healthcare services, clinicians, technologists, designers, and management engineers to stimulate and promote an active lifestyle and prevent health risks among the over-60 population in Lecco and its province.

Active Healthy Aging initiatives, such as the Walking Groups coordinated by local healthcare services, are already active in the Lecco area. This personalized coaching platform aims to leverage these initiatives for prevention and treatment purposes. Its objectives are:

* Creating a user-friendly technological tool for local healthcare services/clinical organizations for projects encouraging physical activity as a driver of lifestyle-based prevention;
* Test this digital therapeutic practice (with a clinical study) on a cohort of 200 individuals to validate its usability, adherence and preliminary efficacy.

The main questions it aims to answer are:

Will a Digital Therapeutics (DTx) based on Active Lifestyle and balance nutrition promotion be adopted and used in an elderly propulation?

What outcomes in health scores will Active3-WP2 platform achieve in physical, metabolic and cognitive domains?

Researchers will compare the use of the proposed DTxA to a contrl gropu receiving a standard educational program.

Participants will:

* receive the Active3-WP2 platform (App+ Wearable)
* participate in health screenings at month 0, month 6 and month 12.

DETAILED DESCRIPTION:
The UN has declared the period 2021-2030 the decade of healthy ageing, based on epidemiological data that show a rapid increase in the elderly population not only in developed countries, but also in middle- and low-income countries.

In this context, the demographic evolution of Italian society over the last twenty years, together with the increase in life expectancy obtained thanks to progress in prevention and treatment approaches, makes the share of the over-60 population increasingly relevant. This population group is heterogeneous but has a significant component of individuals still in work or with good personal and social functioning, although often suffering from one or more chronic diseases or presenting risk factors for future acute or chronic pathological events.

Numerous pieces of evidence confirm that the adoption of healthy lifestyles, with regular physical activity and proper nutrition, is able to have a favorable impact in terms of reducing the risk of morbid events in the neurological and cardiovascular fields through the modification of parameters that are related to these risks. Among these, a particularly important role is played by the body mass index and systolic and diastolic blood pressure values, as well as glycemic and lipid control levels.

In addition to physical activity and diet, other parameters such as satisfactory social interaction are also able to positively influence the so-called healthy ageing, with the consequent cost reductions due to the lower incidence and impact of acute and chronic diseases.

Several studies suggest that the active involvement of recipients of interventions aimed at changing lifestyle habits is a key factor in determining the success of such interventions.

In this line of research, the increasing diffusion of basic digital skills - digital literacy - even in over-60 population groups allows us to believe that people can take advantage of m-coaching approaches with advantage.

However, the adherence to and effectiveness of empowerment models of this nature depends on multiple factors and must be the subject of field trials in sociodemographic contexts in which its possible application on a large scale is expected.

A Spanish multicenter randomized controlled trial has shown a positive short-term effect (3 months) on physical activity and adherence to a Mediterranean diet thanks to the use of an ad hoc app. However, the population to which the intervention was addressed had an average age of 50 years.

In WP2 of the Emblematico Maggiore Active3 - Everyone, Everywhere, Everyday project in the Lecco area and co-funded by the CARIPLO Foundation, the Politecnico di Milano in collaboration with partners is developing a coaching App for the promotion of physical activity as a prevention tool for healthy ageing in the 60-80 age group.

The app records steps and heart rate and weekly food diary and provides motivational feedback to get sedentary people to become active (150 minutes of physical activity weekly) and active people to maintain this healthy lifestyle. The measuring device is a non-medical device device (GARMIN VIVOACTIVE5 or FITBIT) and measures steps and speed and heart rate.

The aim of this study is to analyze the impact of this multidimensional approach, including the use of an e-coaching platform to promote healthy ageing, on adherence to the intervention and on the quality of life of individuals over 60, aged between 60 and 80, in the Lecco area.

The WP2 project of ACTIVE is configured as a RANDOMIZED CONTROLLED CLINICAL TRIAL ON THE IMPACT OF A MULTIDIMENSIONAL APPROACH TO THE EMPOWERMENT OF PEOPLE OVER 60 WITH REFERENCE TO THE ADOPTION OF HEALTHY LIFESTYLES that result in a GENERAL PREVENTION with respect to cardiovascular and metabolic risk.

As part of the Active3 Project and in particular in the WP2 action coordinated by the Politecnico di Milano, a clinical trial entitled "Randomized study of promotion of healthy lifestyles through app versus health education in sedentary individuals or participants in walking groups aged between 60 and 80 years is planned". The promoter of the study is the Politecnico di Milano, the main investigator is Prof. Giuseppe Andreoni, assisted by Dr. Andrea Salmaggi and dr. Enrico Frisone of ASST Lecco and Dr. Stefania Bolis and Dr. Irene Savino of ATS Brianza.

The aim of this study is to analyze the impact of a multidimensional approach including the use of an e-coaching platform to the promotion of healthyaging on the adherence to the intervention and on the quality of life of individuals over 60, aged between 60 and 80, in the Lecco area.

Secondary objectives of the study are possible changes in risk factors, such as blood pressure levels, overweight and glycemic and lipid control levels, as well as any changes in the neuropsychological profile in terms of cognitive performance.

Clinical validation will be carried out on 200 healthy subjects in the 60-80 age group recruited from among participants in walking groups (active) or learners of the University of the Third Age (sedentary) who will adhere on a voluntary basis and upon signing the informed consent to which they will be randomized into 2 groups (intervention and control).

The recruitment will be done in collaboration with ATS-BRIANZA and the tests will be carried out in collaboration with ASST-Lecco (blood and psychological tests), CNR and Villa Beretta (physical and physiological tests).

It is planned to recruit a group of 100 individuals consisting of people already participating in the walking groups coordinated by ATS in the Lecco area, and 100 sedentary people. Individuals will be followed for 12 months and parameters related to primary and secondary outcomes will be monitored before the start of the pathway and at the intermediate (6M) and final time at 12 months.

* Group A1: 50 individuals belonging to the walking groups (Annone, Montevecchia, Lecco) to be administered APP and wearables for 12 months
* Group A2: 50 individuals belonging to the walking groups (Annone, Montevecchia, Lecco) who are NOT administered APPs and wearables for 12 months. (control group)
* Group B1: 50 sedentary individuals from the Municipalities of Annone, Montevecchia, Lecco to whom APPs and wearables are administered.
* Group B2. 50 sedentary individuals preferably from the Municipalities of Annone, Montevecchia, Lecco not to whom APPs and wearables should not be administered A questionnaire on eating habits, BMI assessment, blood pressure values, heart rate, SIX-MINUTE-WALKING TEST, SF-36 scale for quality of life and neuropsychological tests, blood sampling for blood glucose, glycated hemoglobin and cholesterol (total and LDL) will be administered in all participants in enrollment.

The battery of neuropsychological tests administered includes the MMSE and specific tests for different cognitive domains, such as the digit span test, the 15-word list, copy and recall of figures, Raven matrices, attentional matrices, Boston naming test, Trail making test and Wisconsin test short version.

The usability assessment will be carried out with SUS and TAM questionnaires. The data will not be used for medical decisions but only to calculate risk indices: FINDRISC and SCORE2.

Within group A and group B participants will be randomized based on gender, age, and BMI.

The APP will be fed by the data available at baseline with the aim of providing personalized goals, both with regard to the suggested changes in eating habits and with regard to the type and extent of physical exercise required-proposed. The objectives will be given by the APP on a weekly basis.

The wearable provides information on active time, number of steps, distance traveled, heart rate.

A week of physical activity parameters will be measured at the beginning of the trial, based on the individual results that emerged in this monitoring, the APP will set differentiated objectives.

The OUTLINE of the OBJECTIVES BY CATEGORIES AND AGE GROUPS is as follows:

From sedentary to active T0-T6months

* 60-70 years > 3000-4000 daily steps and 90 minutes of physical activity
* 70-75 years > 2100-3500 daily steps and 75 minutes of physical activity
* 75-80 years > 1800-2800 daily steps and 70 minutes of physical activity Sedentary to active T6-T12months
* 60-70 years > 6000-8000 daily steps and 150 minutes of physical activity
* 70-75 years > 4500-7500 daily steps and 130 minutes of physical activity
* 75-80 years > 4000-7000 daily steps and 120 minutes of physical activity Active to trained T0-T6months
* 60-70 years > 6000-8000 daily steps and 200 minutes of physical activity
* 70-75 years > 5500 -7500 daily steps and 180 minutes of physical activity
* 75-80 years > 5000 -7000 daily steps and 150 minutes of physical activity Active to trained T6-T12months
* 60-70 years > 8000-10000 daily steps and 300 minutes of physical activity
* 70-75 years > 7500-9000 daily steps and 250 minutes of physical activity
* 75-80 years > 7000-8500 daily steps and 200 minutes of physical activity

Physical activity is always considered as "moderate"

All participants will be provided with information leaflets upon enrollment in the study with guidance on recommended practices for healthy living, particularly with regard to diet and physical activity.

All individuals will be tested with the following initial, mid-term, and final screening scheme:

1. at month 0 (= at recruitment): all tests;
2. at month 6 (excluding neuropsychological tests);
3. at month 12); all tests.

The ACTIVE3 application, developed for the Android and iOS platforms, is the software with which participants interact with the Active project.

The application is divided into four main parts:

* Motion data
* Walking Group and activities
* Rewards
* Suggestions (nutrition and activity).
* Profile

The App is connected via SpikeAPI to a Garmin VivoActive 5 wearable device. Through this software library, the application is able to record all movement and physical activity data measured through the wearable device. The data collected in this way is stored in a cloud database (Google Firebase cloud) so that it can be analyzed at the end of the clinical study and at the same time be used for the generation of rewards and rankings. The data recorded are:

* Number of daily steps
* Daily moderate active minutes
* Daily vigorous active minutes
* Daily Idle Minutes
* Distance traveled
* HR
* HR at rest The Walking Group and activities part allows you to view the routes and the scheduling of your walking group. The app is therefore also proposed as a means of communicating the calendar of events with participants, confirming attendance, viewing routes and allowing, through GPS, to follow the routes.

Through the data collection of wearables, and based on specific objectives that have been set by clinical partners (based on gender, age and health/activity status), the user receives rewards that can be used in stores (participating in the initiative) to purchase physical goods. In this way, the user is incentivized to achieve the set goals. In addition, the app includes a leaderboard, with which the user can view their placement based on the physical activity they have performed, and receive additional rewards.

The tips section offers the user "health" pills to stay more active and eat healthy. The section works like a real blog, with which you can read these pills. The user can also activate notifications so that they receive a message when a new pill is present in the application.

All data, pills and rewards are stored in the cloud. The database, for privacy reasons, provides for pseudo-anonymization, so all user data are linked to an alphanumeric identifier and are not directly linked to the person. Only by accessing the database of the registry is it possible to link sensitive data to the person himself.

The app, within the profile section, also provides for the compilation of a questionnaire on eating habits based on the Mediterranean diet. The profile section also includes a button requesting account deletion; this option allows you to delete all data from cloud databases as per the specifications required by the GDPR. You can also ask administrators to have a copy of your data.

The data relating to the groups will be analyzed separately, comparing for each group the pre- and post-intervention period data.

Statistical analyses will use parametric and nonparametric tests for continuous variables, while Fischer tests for dichotomous variables will be used.

Evaluation criteria As regards the primary end-point of adherence, a percentage of individuals still active in following the proposed path of 70% in the intervention group is considered satisfactory.

As regards the primary usability end-point, an average SUS score of 75 in the intervention group is considered satisfactory.

As regards the primary end-point of quality of life, an SF-36 is considered satisfactory with a 10% increase pre- and post-intervention.

PRIMARY OBJECTIVES OF THE STUDY

1. Adherence to the proposed route
2. Analysis of the usability of the platform by means of a SUS questionnaire.
3. Assessment of quality of life using the SF-36 scale at times 0, 6 and 12 months in all groups

SECONDARY OBJECTIVES

Preliminary assessment of the clinical efficacy of the behavioral intervention by evaluation of the following indices/parameters:

1. Changes in the BMI - BODY-MASS INDEX
2. CHANGES IN SYSTOLIC AND DIASTOLIC BLOOD PRESSURE LEVELS
3. Changes in the levels of GLYCATED HEMOGLOBIN
4. changes in LDL-CHOLESTEROL levels
5. Changes in SCORES on PSYCHOMETRIC TESTS
6. Changes in SCORE at 6MWT

STATISTICAL ANALYSIS The data relating to adherence will be analyzed by setting the target of 70% of individuals active in the path at 12 months from the start. The vast literature in the field of clinical studies of this type notes that, by way of example, empowerment interventions aimed at lifestyles or the adoption of particular diets are burdened by a drop-out rate of not less than 30%.

Data related to pre- and post-study changes in each subgroup will be analyzed by Student's T-test for paired data. A separate analysis of any drop-outs is also planned in the group, in order to highlight any differences in the pre-trial clinical profile in these compared to the participants who remained active at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 60 and 80 years.

Exclusion Criteria:

* Presence of pathologies, in particular cardio-respiratory diseases, of such severity to prevent the execution of the physical tests and activities promoted by the DTx
* Inability to consent to participate in research.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the DTx | From enrollment to the end of treatment at 12 months
  Adherence to the proposed DTx measured as % of people using the App with at least 1 access per week and 20 minutes per week.
  A percentage of individuals still active in following the proposed path of 70% in the intervention group is considered satisfactory.
Adherence to the DTx | From enrollment to the end of treatment at 12 months
  Adherence to the proposed DTx measured as number of routes taken. Adherence will be measured as average number of routes taken (in the total population).
  A number of walked paths of >25 in the intervention group is considered satisfactory.
Usability | From enrollment to the end of treatment at 12 months
  Usability is considered as satisfaction of use. The satisfaction will be measured by the System Usability Scale (SUS). An average SUS score > 75 in the intervention group is considered satisfactory
Quality of life score | From enrollment to the end of treatment at 12 months.
  Assessment of quality of life using the SF-36 scale at times 0, 6 and 12 months in all groups.
  The SF-36 score provides a 1-100 range score. For each participant will be computed the percentage difference in the score at 6 months and 12 month in comparison to the baseline score.
  The quality of life endpoint (SF-36) is considered satisfactory with a 10% increase pre- and post-intervention (12 months),

SECONDARY OUTCOMES:
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through changes in LDL-CHOLESTEROL levels (mg/dL) in average in the population.
  A reduction of 10 mg/dL will be considered satisfactory.
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through CHANGES IN SYSTOLIC AND DIASTOLIC BLOOD PRESSURE LEVELS (mmHg).
  A reduction > 5 mmHg in systolic blood pressure and 3 mmHg in diastolic blood pressure is considered satisfactory.
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through Changes in the levels of GLYCATED HEMOGLOBIN (%) A reduction of 0,4% will be considered satisfactory.
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through Changes in the BMI - BODY-MASS INDEX (kg/m^2) A reduction of 0.2 kg/m^2 of BMI is considered satisfactory.
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through Changes in SCORES on PSYCHOMETRIC TESTS (a.u.) for MMSE.
  An average increase of 0.5 points in the population will be considered satisfactory.
  Legend:
  a.u- = arbitrary unit
Preliminary assessment of the clinical efficacy of the behavioral intervention | From enrollment to the end of treatment at 12 months
  The Preliminary assessment of the clinical efficacy of the behavioral intervention will be done through the walked distance during the 6MWT (m) The rate of 75% of subjects in the intervention population who will be walking in the expected range defined by Duncan et al. (2015) will be considered satisfactory.
  * Duncan, M.J.; Mota, J.; Carvalho, J.; Nevill, A.M. An Evaluation of Prediction Equations for the 6 Minute Walk Test in Healthy European Adults Aged 50-85 Years. PLoS ONE 2015, 10(9): e0139629. doi:10.1371/journal.pone.0139629.

CONTACTS AND LOCATIONS:
Locations (1):
- Politecnico di Milano - Polo Territoriale di Lecco, Lecco, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No
Privacy issues